CLINICAL TRIAL: NCT07157735
Title: Anti-inflammatory Intervention With Dapansutrile (OLT1177®) for Parkinson's Disease Modification (DAPA-PD): A Randomised Double-Blind, Placebo-Controlled Phase II Trial
Brief Title: A Trial to Test the Use of Dapansutrile, an Anti-inflammatory Medication, in People With Parkinson's Disease
Acronym: DAPA-PD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); Olatec Therapeutics LLC (Industry); Cure Parkinson's (Other); Van Andel Research Institute (Other)
Responsible Party: Principal Investigator, Caroline Williams-Gray, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCTU0443; 348480; 1010807 (Other: Integrated Research Application System)
Record Dates: First submitted 2025-05-15; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Dapansutrile; Neurodegeneration; Neuroinflammation; Inflammation; NLRP3 inflammasome
MeSH Terms: conditions — Parkinson Disease; Nerve Degeneration; Neuroinflammatory Diseases; Inflammation | interventions — dapansutrile

STUDY DESIGN:
Intervention Model Description: Optional open-label phase after 6 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator and outcomes assessor will remain blinded until the end of the open label phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research (Active Comparator)
  Interventions: Drug: dapansutrile
- Control (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dapansutrile — Dapansutrile tablets administered for 26 weeks, starting at 1,000 mg daily (500 mg twice daily) for 4 weeks, escalated to 2,000 mg daily (1,000 mg twice daily) thereafter.
  Arms: Research
Drug: placebo — Matched placebo tablets administered for 26 weeks, admistered as per the active treatment.
  Arms: Control

SUMMARY:
In Parkinson's disease (PD), there is inflammation in the brain, the gut and the blood, which is thought to contribute to the development and progression of the disease. The Nod-like receptor (NLR) family pyrin domain containing 3 (NLRP3) inflammasome is a complex of proteins which plays a critical role in mediating inflammation, and there is growing evidence from laboratory research that the inflammasome plays a role in Parkinson's disease.

Dapansutrile is a new drug which has a highly specific effect on the NLRP3 inflammasome. In animal models, dapansutrile can protect against inflammation in the brain and prevent loss of dopamine cells. Initial 'in human' studies have indicated that this drug can effectively reduce inflammation without causing significant side effects.

The goal of this clinical trial is to test whether dapansutrile might be a useful treatment for Parkinson's disease. The main questions it aims to answer are:

1. is dapansutrile safe and well-tolerated in people with Parkinson's?
2. does dapansutrile reduce inflammation in the brain, cerebrospinal fluid (CSF) and blood? Changes in clinical symptoms will also be measured over the course of the trial.

Researchers will compare dapansutrile to a placebo (a look-alike substance that contains no drug) to see whether it is safe and what effects it has on inflammation and on clinical symptoms.

Participants will be asked to take dapansutrile or a placebo every day for 6 months. Following this, all participants will be given the option to take dapansutrile every day for an additional 6 months. Participants will visit the study centre regularly throughout the trial for check-ups and blood tests. They will have a brain scan before starting treatment and again after 5-6 months. They will also be asked to have a lumbar puncture at the beginning of the trial, after 6 months of treatment and after 12 months of treatment.

DETAILED DESCRIPTION:
DAPA-PD is a randomised double-blind, placebo-controlled phase II trial investigating the safety and tolerability of dapansutrile (OLT1177), an NLRP3 inhibitor, in people with early PD (Hoehn and Yahr stage ≤2, disease duration ≤5 years) who have evidence of peripheral inflammation (high sensitivity C-reactive protein [hsCRP] >1) as an adjunct to dopaminergic therapies. 36 participants will be recruited at a single site and treated with either dapansutrile (1000mg twice daily) or placebo in a 2:1 ratio for a duration of 6 months. This randomised placebo-controlled phase of the trial will be followed by an optional 6-month open label phase, where all participants will receive the active drug. The primary endpoint will be the safety and tolerability of dapansutrile over the 6-month placebo-controlled phase.

Safety data will be collected throughout both phases of the trial, through venous blood sampling, electrocardiograms and clinical assessments. The trial will assess treatment efficacy on peripheral and central inflammation, using biomarkers in blood and CSF, and translocator protein (TSPO) positron emission tomography (PET) brain imaging. Pharmacokinetics of the drug will also be evaluated. Additionally, clinical outcomes, including motor and cognitive progression, will be assessed throughout.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial, the potential participant must:

* Have given written informed consent to participate.
* Be aged between 50 and 80 years (inclusive) at the time of the screening visit.
* Be a fluent English speaker.
* Have a diagnosis of clinically established early PD according to the Movement Disorder Society Criteria for Clinically Established Early Parkinson's Disease.
* Have a disease duration of less than 5 years at the time of screening visit.
* Have early-stage PD, defined as Hoehn and Yahr stage ≤2.
* Be PD drug naïve or be receiving a stable dose of dopaminergic therapy for at least 3 months prior to screening visit, or between screening and baseline.
* Have hsCRP > 1 mg/L at screening visit.
* Have adequate organ function, as defined below (to be rechecked prior to baseline/investigational medicinal product [IMP] initiation if >42 days from screening visit): Haemoglobin ≥ 110 g/L; Platelet count ≥ 130 × 109/L; Neutrophil count ≥ 1.5 × 109/L; Renal function: estimated glomerular filtration rate (eGFR) >45 mL/min/1.73m2; Hepatic function: alanine aminotransferase (ALT) and bilirubin < 1.5 times the institutional upper limit of normal; Thyroid stimulating hormone (TSH) within normal range; Corrected calcium ≤ institutional upper limit of normal; Alkaline phosphatase (ALP) < 1.5 times the institutional upper limit of normal

Exclusion Criteria:

The presence of any of the following will preclude inclusion:

* Low affinity binder for TSPO ligands based on genotyping for single nucleotide polymorphism (SNP) rs6971.
* Any use of immunomodulatory drugs or biologic agents (such as azathioprine, mycophenolate, methotrexate, ciclosporin, cyclophosphamide etc.) within 12 months prior to screening visit, or between screening and baseline.
* Any previous use of rituximab or alemtuzumab at any time.
* Treatment with oral corticosteroids for greater than 2 weeks within 12 months prior to screening visit, or any oral or injected steroid use within 3 months prior to screening visit, or between screening and baseline.
* Regular use of non-steroidal anti-inflammatory drugs (NSAIDs) - including aspirin > 75 mg, naproxen, ibuprofen and meloxicam - on more than 2 days per week.
* Known inflammatory or autoimmune disease.
* Chronic or latent infection.
* Severe infection requiring the use of parenteral antimicrobial agents within 2 months prior to screening visit, or between screening and baseline.
* Skin, solid organ or haematological malignancy within the 5 years prior to screening visit, or between screening and baseline.
* The inability to take or swallow oral medication.
* Parkinson's Disease Dementia according to Movement Disorder Society (MDS) PD Dementia criteria.
* A known genetic mutation associated with PD.
* A positive test for human immunodeficiency virus (HIV), hepatitis B (HBV)/C (HCV) or syphilis.
* Chronic liver disease.
* Any concurrent medical or psychiatric condition or disease that is likely to interfere with the trial procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this trial.
* Women of childbearing potential - female participants must be surgically sterile or be post-menopausal. (A post-menopausal state is defined as no menses for 12 months without an alternative medical cause).
* Male participants must be surgically sterile or must agree to use effective contraception during the period of therapy and for 6 months after the last dose of the trial treatment.
* Known hypersensitivity to dapansutrile or its excipients.
* Received an investigational drug or used an invasive investigational medical device within 12 weeks before the screening assessment, or is currently enrolled in another interventional investigational trial. Participants currently enrolled in other observational studies may be recruited.
* Contraindications to PET-magnetic resonance imaging (MRI) scanning including metal implants, claustrophobia or inability to lie flat for 90 minutes.
* Concomitant treatment with any medications that could interfere with [18F] DPA-714 binding (e.g., benzodiazepines).
* Current use of any drugs of abuse or average alcohol intake of >21units per week over the last 3 months.
* Any other significant disease, disability or investigation result which, in the opinion of the Chief Investigator (CI), may either put the participant at risk, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events (AEs) recorded during the 6-month double-blind period | Assessed at screening, baseline, day 1, and weeks 2, 4, 6, 12, 18, 23 and 26.
  Adverse events are recorded from the point of participant informed consent and at every trial visit

SECONDARY OUTCOMES:
Change in [¹⁸F]-DPA-714 PET non-displaceable binding potential in subcortical and cortical regions of interest | Between baseline and week 23
  Measured using PET- magnetic resonance (MR) brain imaging with [¹⁸F]-DPA-714, a TSPO ligand.
Change in concentration of C-reactive protein (CRP) in blood | Over 6 months of treatment, measured at day 1, and weeks 6, 18 and 26.
Change in concentration of interleukin (IL)-1β in blood | Over 6 months of treatment, measured at day 1, and weeks 6, 18 and 26.
Change in concentration of interferon (IFN)-γ in blood | Over 6 months of treatment, measured at day 1, and weeks 6, 18 and 26.
Change in concentration of IL-18 in blood | Over 6 months of treatment, measured at day 1, and weeks 6, 18 and 26.
Change in concentration of IL-6 in blood | Over 6 months of treatment, measured at day 1, and weeks 6, 18 and 26.
Change in concentration of tumour necrosis factor (TNF)-α in blood | Over 6 months of treatment, measured at day 1, and weeks 6, 18 and 26.
Change in concentration of apoptosis-associated speck-like protein containing a CARD (ASC) specks in blood | Over 6 months of treatment, measured at day 1, and weeks 6, 18 and 26.
Change in concentration of CRP in CSF | Over 6 months of treatment, measured at baseline and week 26.
Change in concentration of IL-1β in CSF | Over 6 months of treatment, measured at baseline and week 26.
Change in concentration of IL-18 in CSF | Over 6 months of treatment, measured at baseline and week 26.
Change in concentration of IL-6 in CSF | Over 6 months of treatment, measured at baseline and week 26.
Change in concentration of TNF-α in CSF | Over 6 months of treatment, measured at baseline and week 26.
Change in concentration of ASC specks in CSF | Over 6 months of treatment, measured at baseline and week 26.
Pharmacokinetics as measured by changes in plasma and CSF dapansutrile concentrations | Between baseline and end of treatment; measured in the blood at day 1, and weeks 6, 18 and 26; and measured in CSF at baseline and week 26.

OTHER OUTCOMES:
Number of AEs recorded | During the 6-month open-label period
Change in Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III | Between baseline and 6 months, and over 12 months (if performed)
  MDS-UPDRS part III will be used to measure the change in motor examination. Scoring ranges from 0 to 132, with a higher score indicating more severe motor impairment.
Change in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) gait/axial score | Between baseline and 6 months, and over 12 months (if performed).
  This score is a sum of the points from the following sections of MDS-UPDRS part III: speech, facial expression, rising from a chair, gait, postural stability, posture, and body bradykinesia. Scoring ranges from 0 to 28. A higher score is more severe.
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I | Between baseline and 6 months, and over 12 months (if performed)
  Part I of the MDS-UPDRS assesses Non-Motor Aspects of Experiences of Daily Living (nM-EDL). Scoring ranges from 0 to 52, with higher scores indicating more severe symptoms.
Change in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part II | Between baseline and 6 months, and over 12 months (if performed).
  Part II of the MDS-UPDRS assesses Motor Aspects of Experiences of Daily Living (M-EDL). Scoring ranges from 0 to 52, with higher scores indicating more severe symptoms.
Change in Addenbrooke's Cognitive Examination-III (ACE-III) | Between baseline and 6 months, and over 12 months (if performed)
  ACE-III is a global cognitive assessment tool. Scores range from 0 to 100, with higher scores indicating better cognitive functioning.
Change in Movement Disorder Society-Non-Motor Rating Scale (MDS-NMS) | Between baseline and 6 months, and over 12 months (if performed)
  MDS-NMS measures the burden of non-motor symptoms, including non-motor fluctuations in Parkinson's disease. Scores range from 0 to 180 with higher scores indicating a greater symptom burden.
Change in Gastrointestinal Dysfunction Scale for Parkinson's Disease (GIDS-PD) | Between baseline and 6 months, and over 12 months (if performed)
  GIDS-PD is a patient-reported outcome measure of gastrointestinal symptoms in Parkinson's disease. Scores range from 1 to 108, with a higher score representing a greater number and/or severity of gastrointestinal symptoms.
Geriatric Depression Scale-30 (GDS-30) | Between baseline and 6 months, and over 12 months (if performed)
  GDS-30 is a patient-reported outcome measure of depression. Scores range from 0 to 30, with a higher score indicating greater severity of depression.
Parkinson's Disease Questionnaire-39 (PDQ-39) | Between baseline and 6 months, and over 12 months (if performed).
  PDQ-39 is a patient-reported outcome measure of quality of life in Parkinson's disease. Scores range from 0 to 100 with a higher score indicating greater functional impairment and lower quality of life .
Changes in other inflammatory markers related to inflammasome activation in the blood and CSF, which are deemed relevant by the investigators | Between baseline and 6 months, and over 12 months (if performed)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Williams-Gray, BMBCh MA(Cantab) FRCP PhD, Principal Investigator — University of Cambridge
Locations (1):
- John Van Geest Centre for Brain Repair, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided